CLINICAL TRIAL: NCT01931501
Title: An Open Label, Randomized, Two-Period, Two-Treatment, Crossover, Single-Dose Bioequivalence Study of Montelukast Sodium Chewable Tablets 5mg [Test Formulation, Torrent Pharmaceutical Limited., India] Versus Singulair® (Montelukast Sodium) Chewable Tablets 5mg [Reference Formulation, Merck & Co., Inc. USA] in Healthy Human Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Ltd.'s Montelukast Sodium Chewable Tablets 5mg Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized
Other Study IDs: PK-07-117
Record Dates: First submitted 2013-08-21; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
MeSH Terms: interventions — montelukast

INTERVENTIONS:
Drug: Torrent's Montelukast Sodium Chewable Tablets 5mg
Drug: Singulair® (Montelukast Sodium) Chewable Tablets 5mg

SUMMARY:
Objective:

Primary objective of the present study was to compare the single dose bioavailability of Torrent's Montelukast Sodium chewable 5 mg tablet and Innovator's(Merck)Singulair chewable 5 mg tablet. Dosing periods were separated by a washout period during fasted study.

Study Design:

Open-Label, Randomised, two Period, two treatment, Crossover, Single-Dose Bioequivalence Study

ELIGIBILITY:
Inclusion Criteria:

The volunteers were included in the study based on the following criteria:

Sex: male.

* Age: 18 - 45 years.
* Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day

Exclusion Criteria:

The volunteers were excluded from the study based on the following criteria:

* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute.
* Oral temperature less than 95°P or more than 98.6°P.
* Respiratory rate less than 12/minute or more than 20/minute
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* History of alcohol or drug abuse
* Positive breath alcohol test
* Recent history of kidney or liver dysfunction.
* History of consumption of prescribed medication since last 14 days or OTC medication since last 07 days before beginning of the study.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of heart failure.
* HIV, HCV, HBsAg positive volunteers.
* Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, - - - Cocaine positive volunteers based on urine test.
* Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
* Administration of any study drug in the period 0 to 3 months before entry to the study.
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* History of pre-existing bleeding disorder.
* Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
* Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
bioequivalence based on Composite of Pharmacokinetics | plasma samples were obtained from blood drawn at Pre-dose and 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 10.00, 12.00, 14.00 and 24.00 hours after dose administration.
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio Evaluation Centre, Torrent Pharmaceuticals Ltd., Village Bhat, Gandhinagar, Gujarat, India